CLINICAL TRIAL: NCT06025266
Title: Investigation of the Acute Effect of Foot Extrinsic Muscle Fatigue on Viscoelastic Properties of the Plantar Fascia and Achilles Tendon
Brief Title: Investigation of the Effect of Foot Muscle Fatigue on the Foot Sole and Tendon Structural Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simge Dönmez (Other)
Responsible Party: Sponsor-Investigator, Simge Dönmez, Physiotherapist, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 11-959
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Healthy Participants
Keywords: viscoelastic properties; MyotonPRO; fatigue; plantar fascia; Achilles tendon
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: The same 19 people were seen 3 times to evaluate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unilateral Heel Raise (Experimental): Muscle fatigue was created by exercise consisting of a combination of repetitive plantar flexion and dorsiflexion movements performed during the entire range of motion of the ankle at the frequency of movement determined by the metronome on one step.
  Interventions: Device: Evaluation of Viscoelastic and mechanical properties with MyotonPRO
- Closed Chain Resisted Foot Adduction (Experimental): The exercise was performed on the designed wooden assembly. The device was used to maintain the neutral position of the subtalar joint, stabilize the lateral and medial malleoli, and prevent compensation with the knee and hip joints. Individuals were seated with the knee flexed approximately 80 degrees and separated from the other extremity by the length of the forearm, and the contralateral knee was stabilized with the ipsilateral hand. The foot was brought from the abduction position to the adduction position and the heel was not lifted from the ground throughout the movement. The exercise was performed using a green elastic band.The movement was performed in sets of 50 concentric/eccentric contractions. A rest period of 10 seconds was added between each set.
  Interventions: Device: Evaluation of Viscoelastic and mechanical properties with MyotonPRO
- Combined Exercise (Experimental): Unilateral Heel Raise and Closed Chain Resisted Foot Adduction exercises were performed sequentially.
  Interventions: Device: Evaluation of Viscoelastic and mechanical properties with MyotonPRO

INTERVENTIONS:
Device: Evaluation of Viscoelastic and mechanical properties with MyotonPRO — MyotonPro™, a handheld, non-invasive and painless device, is used for non-invasive measurement of the biomechanical and viscoelastic properties of soft biological tissues such as superficial skeletal muscles, fascia, tendons and ligaments. The properties of the structures can be measured from different regions during complete rest or contraction.

SUMMARY:
In healthy individuals, fatigue in the foot muscles increases the load and stress on the feet. The extrinsic muscles of the foot, which investigators aimed to create fatigue in this study, are closely related anatomically and functionally to the plantar fascia and Achilles tendon. Considering that fatigue or weakness of the foot extrinsic muscles is an important risk factor for foot-ankle pathologies, it is important to reveal the relationship with the plantar fascia and Achilles tendon in healthy sedentary individuals and to determine mechanical properties of the feet of the participants to prevent possible foot injuries. Therefore, the aim of this study is to show the acute effects of fatigue in the extrinsic muscles of the foot on the viscoelastic properties of the plantar fascia and Achilles tendon. The study was completed with 19 people who met the inclusion criteria. Before starting the study, the dominant foot of the participants was determined, physical activity level was determined, foot posture index and foot posture were evaluated, navicular height and fall distance of the foot were measured, m.gastrocnemius shortness was measured with the Silfverskiöld test, flexibility was evaluated with a baseline sitting bench, tendon and fascia measurements were made with the MyotonPRO device. After the measurements, the participant was trained to perform the heel raise exercise. When the exercise was completed, the participant's foot Myoton measurements were repeated. One week later, pre-exercise Myoton measurement was performed, then the participant was trained for the foot adduction exercise. When the exercise was completed, the participant's foot Myotone measurements were repeated. In another week, pre-exercise Myotone measurement was performed, then heel raising and foot adduction exercises were performed sequentially. When the exercise was completed, the participant's foot Myoton measurements were repeated.

DETAILED DESCRIPTION:
This study was carried out on healthy, sedentary male individuals between the ages of 18-35. In the power analysis to estimate the sample size, Usgu et al. (2020), it was determined that there should be a minimum of 17 observations in each group, with a statistical power level of 82.2% and a significance level of 5%. The study was completed in 3 groups in line with the selected exercises. Firstly, 42 young individuals were included in the study. However, after the preliminary evaluation, 23 individuals who did not meet the inclusion criteria and did not provide continuity to the study were excluded from the study. This study was completed with 19 healthy male individuals with a mean age of 21.37(SD 2.21) years.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study voluntarily
* Being a healthy, sedentary male individual between the ages of 18 and 35
* Being in categories 1 and 2 according to the International Physical Activity Survey (UFAA)
* Having a normal Body Mass Index (BMI) (18.5 kg/m2 ≤ BMI ≤24.9 kg/m2)
* Having a neutral foot posture (<6 points in the Foot Posture Index)

Exclusion Criteria:

* Refusing to participate in the study or wanting to leave the study
* Having a history of previous surgery in the lower extremity
* Being diagnosed with a musculoskeletal disease
* Having any chronic disease (hypertension, diabetes, cardiovascular disease, osteoporosis, rheumatism, etc.)
* Having a skin lesion in the area to be measured
* Significant weakness in the lower extremity gross muscle test
* Any limitation in the normal range of motion of the lower extremity
* Having any deformity in the foot (pes planus, pes cavus, hallux valgus)
* Navicular drop distance ≥10 mm
* Limitation in the range of motion of the 1st metatarsophalangeal joint (hallux rigidus-limitus)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males were included, as sex hormones could affect the structural properties of soft tissues such as muscle and fascia.
Enrollment: 19 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Biomechanical and viscoelastic properties of tissue | 3 weeks
  Biomechanical and viscoelastic properties of AT and PF were performed using MyotonPro™ (Myoton AS, Tallinn, Estonia) device. Before and immediately after the application of the fatigue protocol, AT and PF measurements were made separately with the MyotonPro™ device. The measurement points determined for AT and PF of individuals during rest were marked with a medical marker pen (16). The measurement points of each person and their distances to the anatomical points were measured with the help of a tape measure and recorded in their files to find the same point again. During the measurement, the probe of the device was adjusted to pulse once into the skin with a force of 0.4 N and for 15 ms. During the test, the tip of the MyotonPro™ device was placed perpendicular to the marked area and gently pressed against the skin at a depth of 3 mm until the green light came on.

SECONDARY OUTCOMES:
Identifying the Dominant Foot | 1 day
  The dominant foot was determined using the ball-kicking method. While the individual was standing, a ball was placed in the middle of both feet and the individual was asked to hit the ball with his foot. The extremity on which the individual hit the ball was accepted as dominant.
  The dominant foot was determined using the ball-kicking method. While the individual was standing, a ball was placed in the middle of both feet and the individual was asked to hit the ball with his foot. The extremity on which the individual hit the ball was accepted as dominant.
Physical Activity Level | 1 day
  The physical activity level of the individuals was evaluated with the International Physical Activity Questionnaire (IPAQ)-Short Form. This scale, whose short form consists of 7 items, provides information about the time spent during the activity by classifying the activity according to the differences in intensity level. Total Physical Activity Score; The vigorous and moderate physical activity and walking times of the participants in the last 7 days were calculated with the formulas by multiplying the minutes, the number of days and the MET-minute score appropriate for the physical activity performed (MET (Metabolic Equivalent of Task)-min/week). According to the questionnaire, physical activity levels are those who are not physically active (<600 MET-min/week), low physical activity level (600-3000 MET-min/week) and adequate physical activity level (beneficial for health) (> 3000 MET-min/week).
Sit-Reach Test | 1 day
  In particular, a sit-reach bench (Baseline®, Cooper Institute/YMCA, AAHPERD, New York, USA) was used to measure the flexibility of the lower back and hamstring muscles. Subjects were asked to contact a standard sit-and-reach bench in a sitting position, with their backs against the wall and their knees in full extension, with the soles of their feet flat on the box. Then, individuals were asked to reach forward as far as possible by pushing the device apparatus with their fingertips without lifting their knees, with their palms facing down. Measurements were repeated 3 times and the average of the values was recorded.
Silfverskiold Test | 1 day
  The muscle shortness assessment of the individuals regarding M. Gastrocnemius was performed on both ankles while in the supine position using the Silfverskiold method and universal goniometer. While the knee joint was in full extension and 90° flexion, and the subtalar joint was in the neutral position, the dorsiflexion of the ankle was passively performed by the assessor, and the fixed arm of the universal goniometer was measured on the fibula shaft and the mobile arm was placed on the fifth metatarsal shaft. The resulting angles were recorded in degrees.
Navicular Height | 1 day
  The navicular height was defined as the distance of the navicular tubercle to the ground when the individual was standing in a relaxed position. In our study; Subjects were asked to stand in a comfortable position for navicular height assessment. The medial protrusion of the tuberosity of the navicular was detected and marked by palpation, and the distance between this point and the ground was measured using a millimetric ruler. The result is recorded in millimeters
Navicular Drop Distance | 1 day
  Before the measurement, the medial protrusion of the tuberosity of the navicular was detected and marked by palpation. The height of the navicular tubercle was determined with the help of a millimetric ruler placed on the medial part of the foot while the individuals were sitting in a chair with the soles of their feet touching the ground and the hips and knees flexed to 90°. Individuals were asked to stand up and the height of the navicular tubercle was determined again. The amount of change was determined with the help of a ruler and recorded. Each measurement was repeated 3 times and the average value was recorded in millimeters.
Evaluation of Foot Posture | 1 day
  Foot Posture Index-6 was used to evaluate foot posture. During the evaluation, the subjects were asked to stand in a way that was comfortable, without moving. Test; It was performed by the physiotherapist based on observation and palpation while the individual was in a static and comfortable standing position. The index consists of 6 items in total, 3 items in the forefoot and 3 items in the hindfoot. In the study; Evaluations were made bilaterally based on observation and palpation from the posterior, medial, lateral and anterior aspects.
Evaluation of Fatigue | 3 weeks
  The level of fatigue perceived by the individuals during the study was evaluated with the "Borg Fatigue Scale" immediately after completing the fatigue protocol exercises. Developed by Borg, this scale has 10 levels in its modified form, and the category ratio scale consists of definitions corresponding to certain numbers. The participant was asked to score the perceived fatigue between 0 (not at all) and 10 (very very hard).

CONTACTS AND LOCATIONS:
Overall Officials: Simge Dönmez, Principal Investigator — Kütahya Health Sciences University; Fatmagül Varol, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No